CLINICAL TRIAL: NCT05430828
Title: Multicenter Study on the Evaluation of Adherence, Persistence and Efficacy of Treatment With PCSK9 Inhibitors in Italy
Brief Title: Evaluation of Adherence, Persistence and Efficacy of Treatment With PCSK9 Inhibitors in Italy
Acronym: AT-TARGET-IT
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Other Study IDs: 264/20
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab; alirocumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Subjects with hyperlipidaemia under PCSK9 inhibitors treatment (Repatha/Praulent).
  Interventions: Drug: Repatha (evolocumab); Praluent (alirocumab)

INTERVENTIONS:
Drug: Repatha (evolocumab); Praluent (alirocumab) — Dosage form: Injection

SUMMARY:
Evaluation of adherence, persistence and efficacy of treatment with PCSK9 inhibitors in a real-life Italian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients under PCSK9 inhibitor treatment.

Exclusion Criteria:

* Age < 18 years o > 80 years;
* Patients who refuse to participate and to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients from Italy, who have received PCSK9 inhibitor as part of routine clinical management of their hyperlipidaemia for at least 6 months at time of enrollment, based on national reimbursement criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-07 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Description of adherence of treatment with PCSK9 inhibitors in a real-life Italian population. | every 6 months
  Adherence will be assessed in terms of Medical Possession Ratio (MPR) which is defined as the ratio between the treatment units dispensed during the treatment period and the duration of the treatment period itself. MPR will be calculated as overall MPR (mean and median value), MPR by type of prevention (primary and secondary), MPR by type of antiPCSK9 inhibitor (alirocumab vs. evolocumab), MPR by type of background therapy (statin yes, statin no) , MPR by demographic variables (age, sex, geographic origin, basal LDL levels), MPR by type of prescriber (hospital or territorial).
Description of persistence of treatment with PCSK9 inhibitors in a real-life Italian population. | every 6 months
  Persistence will be assessed in terms of therapeutic continuity from the start of treatment to enrollment.
Description of efficacy of treatment with PCSK9 inhibitors in a real-life Italian population. | every 6 months
  Efficacy of treatment will be evaluated as a change in the LDL (deltaLDL) value from the start of treatment (percentage and absolute value). The deltaLDL will be calculated as an overall (mean and median value), by type of prevention (primary and secondary), by type of antiPCSK9 inhibitor (alirocumab vs. evolocumab), by type of basic therapy (statin yes, statin no), by demographic variables (age, sex, geographic origin, basal LDL levels), by type of prescriber (hospital or territorial).

SECONDARY OUTCOMES:
Description of adherence, efficacy and safety of treatment with PCSK9 inhibitors in a real-life Italian population general and divided into subgroups. | every 6 months
  Safety will be evaluated in terms of adverse reactions or intolerance to the drug.

CONTACTS AND LOCATIONS:
Locations (27):
- Italy (27):
  - Ospedali dell'Ovest Vicentino, Arzignano
  - University of Bari Aldo Moro, Bari
  - University of Campania Luigi Vanvitelli, Caserta
  - University Magna Graecia of Catanzaro, Catanzaro
  - Presidio Ospedaliero Maria SS Addolorata, Eboli
  - Policlinico Riuniti Foggia, Foggia
  - Università degli Studi di Genova, Genova
  - Ospedale di Lecce, Lecce
  - Università degli Studi di Messina, Messina
  - Policlinico di Milano Ospedale Maggiore - Fondazione IRCCS Ca' Granda, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AORN dei Colli - Ospedale monaldi, Napoli
  - Federico II University of Naples, Department of Advanced Biomedical Sciences, Napoli
  - Federico II University of Naples, Department of Translational Medical Sciences, Napoli
  - University of Naples Federico II, Department of Clinical Medicine and Surgery, Napoli
  - Azienda Ospedaliero-Universitaria "Maggiore della Carità", Novara
  - Azienda Ospedaliero-Univeristaria di Parma, Parma
  - Presidio Ospedaliero Pescara, Pescara
  - Ospedale di Rivoli, Rivoli
  - Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Policlinico Casilino, Roma
  - Sapienza University of Rome, Roma
  - Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale SS Annunziata A.O.U., Sassari
  - University of Siena, Siena
  - Azienda Ospedaliera Ordine Mauriziano Torino, Torino